CLINICAL TRIAL: NCT04710433
Title: Non-invasive Sacral Nerve Stimulation in Children and Adolescents With Chronic Constipation: a Case-control Study on External Neuromodulatory Treatment
Brief Title: Non-invasive Sacral Nerve Stimulation in Children and Adolescents With Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, Dr. med. Sonja Diez, M.D., Friedrich-Alexander-Universität Erlangen-Nürnberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18_20B1
Record Dates: First submitted 2021-01-08; First posted 2021-01-14 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Chronic Constipation With Overflow; Encopresis With Constipation and Overflow Incontinence; Hirschprung's Disease; Anorectal Malformations
Keywords: Sacral Nerve Stimulation; Neuromodulation
MeSH Terms: conditions — Anorectal Malformations | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive Neuromodulation (Active Comparator): Application of non-invasive sacral nerve stimulation for 12 weeks, at least 8 hours per day.
  Two adhesive electrodes are placed paravertebrally between L1 and L4 and periumbilically, generating an electrical field with a 15 Hz frequency for a duration of 210µs. Stimulation intensity is individually determined to achieve an effective and comfortable stimulation beyond the pain threshold (adjustable amplitude between 0-10mA).
  Medical and behavioral therapy is to be continued as started before intervention.
  Interventions: Device: Non-invasive Neuromodulation
- Medical/behavioral Therapy (Other): Patients receive an optimized conventional treatment for 12 weeks, including lifestyle changes, toilet training and weight-adjusted medication. Conventional medical options include oral laxative medication with polyethyleneglycol or rectal medication with saline enemas in possible combination with a stimulant laxative (glycerin or bisacodyl).
  Interventions: Other: Medical and Behavioral Therapy

INTERVENTIONS:
Device: Non-invasive Neuromodulation — Sacral nerve stimulation via two adhesive electrodes (single current).
  Arms: Non-invasive Neuromodulation
Other: Medical and Behavioral Therapy — Behavioral Therapy consists of toilet training, an active and healthy lifestyle. Doses of medical options are applied weight-adjusted.
  Arms: Medical/behavioral Therapy

SUMMARY:
The purpose of this study is to assess the efficacy of additional neuromodulation for treatment of chronic constipation in pediatric patients

DETAILED DESCRIPTION:
Patients are selected according to the eligibility requirements. After being informed about the study and potential risks of neuromodulation, all included patients and next of kin give written informed consent to the study.

At baseline, patients are classified to one of the two predefined subgroups: either medical and behavioral therapy is extended and optimized or neuromodulatory treatment is started with non-invasive sacral nerve stimulation via single current and two external adhesive electrodes. Within 12 weeks, treatment success is evaluated in routine clinical check-ups (week 4/8/12) and via specialized questionnaires and bowel movement diaries. Quality of life is evaluated at baseline and after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* age between 2-17 years
* informed consent
* chronic constipation according to the ROME IV criteria for more than 3 months with or without encopresis/soiling
* refractory to conventional treatment in a sufficient application (training for bowel movements, lifestyle changes, pelvic floor training)
* exclusion of metabolic, inflammatory and hormonal causes for chronic constipation (such as e.g., celiac disease, cystic fibrosis, hypothyroidism)
* in cases of underlying Hirschsprung's disease: confirmation of diagnosis via rectal biopsies
* in cases of anorectal malformation: post-surgical status

Exclusion Criteria:

* metabolic, inflammatory and hormonal causes for chronic constipation with further therapeutic options
* toxic megacolon or further emergencies, which must be treated surgically
* fractures or substantial differences in the sacral anatomy
* inflammatory bowel disorders
* rectal prolapse
* neuronal malignancies under medical and radiation therapy
* seizures

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Symptoms: Change in defecation frequency | Baseline and 12 weeks after start of therapy
  Defecation frequency is measured by bowel movements per week.
Symptoms: Change in defecation consistency | Baseline and 12 weeks after start of therapy
  Defecation consistency is measured by the Bristol Stool Scale, which classifies stool consistency from 1 (hard consistency) to 7 (fluid consistency).
Symptoms: Change of encopresis/soiling | Baseline and 12 weeks after start of therapy
  Episodes of encopresis/soiling are evaluated per day.
Change in Quality of Life | Baseline and 12 weeks after start of therapy
  The quality of life is classified via the 'Revised Children's Quality of Life Questionnaire' (KINDLR). It consists of 24 5-point Likert-scale items, covering 6 quality of life dimensions: physical well-being, emotional well-being, self-esteem, family, friends and daily functioning (school or nursery school/kindergarten). Items are partially reverse scored and linearly transformed to a 0 to 100 scale according to the manual. Higher scores indicate a better quality of life.

SECONDARY OUTCOMES:
Symptoms: Change of abdominal pain | Baseline and 12 weeks after start of therapy
  Abdominal pain is recorded in episodes per week and its intensity is evaluated via the numeric rating scale (0=no pain, 10=worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Diez, MD, Principal Investigator — Friedrich-Alexander-Universität Erlangen-Nürnberg; Manuel Besendörfer, MD, Principal Investigator — Friedrich-Alexander-Universität Erlangen-Nürnberg
Locations (1):
- Friedrich-Alexander-Universität Erlangen-Nürnberg, Pediatric Surgery, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Besendorfer M, Kohl M, Schellerer V, Carbon R, Diez S. A Pilot Study of Non-invasive Sacral Nerve Stimulation in Treatment of Constipation in Childhood and Adolescence. Front Pediatr. 2020 Apr 16;8:169. doi: 10.3389/fped.2020.00169. eCollection 2020. PMID 32373563